CLINICAL TRIAL: NCT04202302
Title: The Impact of Vaginal Profile During Ovarian Stimulation on the IVF/ICSI Outcome: a Prospective Observational Study
Brief Title: Vaginal Profile in IVF/ICSI and Impact on Clincal Outcome
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University (Other)
Responsible Party: Principal Investigator, Haiyan Lin, Principal Investigator, Sun Yat-Sen Memorial Hospital of Sun Yat-Sen University
Other Study IDs: SYSEC-KY-KS-2019-161
Record Dates: First submitted 2019-12-15; First posted 2019-12-17 (Actual); Last update posted 2019-12-18 (Actual); Status verified 2019-12

CONDITIONS: Vaginal Flora Imbalance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: IVF/ICSI — ovarian stimulation ，vaginal disinfection of flushing

SUMMARY:
Vaginal flora is closely related to female reproductive health. Previous studies have suggested that the composition of the vaginal flora is related to the pregnancy outcomes, and abnormalities in the vaginal flora lead to a decrease in the success rate of IVF. During the IVF treatment, the hormone level changes far exceed the physiological level. What changes will happen to the vaginal flora? Does IVF treatment itself affect the vaginal flora and affect outcomes? This study used prospective cohort study to show the changes in vaginal flora during conventional IVF treatment, providing more evidence for revealing the relationship between vaginal flora and infertility treatment outcomes.

ELIGIBILITY:
Inclusion Criteria:

* 20-40 years old
* BMI<30kg/m2
* First IVF/ICSI cycle (GnRH agonist or antagonist protocol)
* no vaginitis after recruitment
* completion of oocyte retrieval

Exclusion Criteria

* history of RSA
* history of endometriosis
* Immune diseases such as SLE, etc., and the use of immunosuppressive agents, glucocorticoids, etc.
* obvious hydrosalpinx(>2cm in diameter by ultrasound)

Ages: 20 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: The study population is from the infertility patients of reproductive center of Sun Yat-sen Memorial Hospital.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2019-08-06 (Actual); Primary Completion 2020-03 (Estimated); Study Completion 2020-03 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rate | 12.2019-03.2020
  no. of clinical pregnancy / total number of embryo transfer cycles

CONTACTS AND LOCATIONS:
Locations (1):
- Reproductive center of Sun Yat-sen memorial hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: Undecided